CLINICAL TRIAL: NCT01218802
Title: Randomized Placebo-controlled Trial of Rosuvastatin in HIV-Infected Subjects to Modulate Cardiovascular Risk and Inflammation
Brief Title: Use of Rosuvastatin in HIV-Infected Subjects to Modulate Cardiovascular Risks
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); AstraZeneca (Industry)
Responsible Party: Principal Investigator, Grace McComsey, Chief, Peds ID, Rheumatology and Global Health, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1R01NR012642-01 (NIH)
Record Dates: First submitted 2010-10-08; First posted 2010-10-11 (Estimated); Results first posted 2016-03-08 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: HIV Infections; Heart Disease
Keywords: HIV; Heart Disease; Bone Density
MeSH Terms: conditions — HIV Infections; Heart Diseases | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rosuvastatin (Active Comparator): Participants will take Rosuvastatin 10 mg. daily for 96 weeks
  Interventions: Drug: Rosuvastatin 10 mg. daily for 96 weeks
- Sugar Pill placebo (Placebo Comparator): Participants will take a placebo that appears on the exterior to be the same as active drug. They will take one capsule daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rosuvastatin 10 mg. daily for 96 weeks — Participants will take Rosuvastatin 10 mg. daily for 96 weeks.
  Other Names: Crestor
  Arms: Rosuvastatin
Drug: Placebo — participants will take a sugar pill daily for 96 weeks
  Arms: Sugar Pill placebo

SUMMARY:
The hypothesis of this study is that 96 weeks of Rosuvastatin will be safe and effective in decreasing cardiovascular risk and bone loss in the HIV+ population.

DETAILED DESCRIPTION:
While the use of antiretroviral therapy (ART) in recent years has had an impressive impact on mortality and disease progression in HIV-infected patients, nevertheless, cardiovascular disease is a major concern impacting morbidity and mortality in this population.

This study will assess if a potent statin, rosuvastatin, could improve endothelial dysfunction, slow carotid intima media thickness (IMT) progression and bone loss, and decrease inflammation and oxidative stress in HIV-infected ART-treated subjects with good HIV virologic control. The investigators will also see if rosuvastatin will induce beneficial changes in the prevalence of metabolic syndrome and lipid metabolism as well as improve bone turnover markers.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of HIV Disease
* Age > 18 years old
* Receiving a stable ARV regimen for at least the last 12 weeks prior to study entry and cumulative duration of ARV for 12 months
* Fasting LDL cholesterol < 130 mg/dl
* Fasting triglycerides < 300 mg/dL
* hsCRP > 2 mg/L or CD38+DR+/CD8+ > 19%
* If on Vit D replacement therapy, stable regimen for > 3 months prior to study entry

Exclusion Criteria:

* Women who are pregnant or breast feeding
* Any active or chronic inflammatory condition
* Cardiovascular disease
* Current or recent (within 24 weeks of study entry) therapy with omega-3 fatty acids, fibrates, ezetimibe or statins
* Uncontrolled hypothyroidism or hyperthyroidism
* Uncontrolled diabetes
* Use of systemic cancer chemotherapy of immunomodulating agents
* Use of Anabolic agents, growth hormone, growth hormone releasing factor, or any other anabolic agents, except for stable replacement testosterone.
* Use of biphosphonates or other bone therapies
* Any of the following lab findings obtained within 14 days prior to the screening evaluation including the following:

  * AST and/or ALT > 2.5 x ULN
  * Hemoglobin < 9.0 g/dL
  * CK > 3 X ULN
  * Calculated creatinine clearance < 50 mL/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2011-02; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grace McComsey, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals of Cleveland Case Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Derived] El Kamari V, Hileman CO, Gholam PM, Kulkarni M, Funderburg N, McComsey GA. Statin Therapy Does Not Reduce Liver Fat Scores in Patients Receiving Antiretroviral Therapy for HIV Infection. Clin Gastroenterol Hepatol. 2019 Feb;17(3):536-542.e1. doi: 10.1016/j.cgh.2018.05.058. Epub 2018 Jun 14. PMID 29908359
- [Derived] Dirajlal-Fargo S, Webel AR, Longenecker CT, Kinley B, Labbato D, Sattar A, McComsey GA. The effect of physical activity on cardiometabolic health and inflammation in treated HIV infection. Antivir Ther. 2016;21(3):237-45. doi: 10.3851/IMP2998. Epub 2015 Oct 12. PMID 26455521
- [Derived] Hale AT, Longenecker CT, Jiang Y, Debanne SM, Labatto DE, Storer N, Hamik A, McComsey GA. HIV vasculopathy: role of mononuclear cell-associated Kruppel-like factors 2 and 4. AIDS. 2015 Aug 24;29(13):1643-50. doi: 10.1097/QAD.0000000000000756. PMID 26372274
- [Derived] Hileman CO, Dirajlal-Fargo S, Lam SK, Kumar J, Lacher C, Combs GF Jr, McComsey GA. Plasma Selenium Concentrations Are Sufficient and Associated with Protease Inhibitor Use in Treated HIV-Infected Adults. J Nutr. 2015 Oct;145(10):2293-9. doi: 10.3945/jn.115.214577. Epub 2015 Aug 12. PMID 26269240
- [Derived] Erlandson KM, Jiang Y, Debanne SM, McComsey GA. Rosuvastatin Worsens Insulin Resistance in HIV-Infected Adults on Antiretroviral Therapy. Clin Infect Dis. 2015 Nov 15;61(10):1566-72. doi: 10.1093/cid/civ554. Epub 2015 Jul 8. PMID 26157049
- [Derived] Lipshultz HM, Hileman CO, Ahuja S, Funderburg NT, McComsey GA. Anaemia is associated with monocyte activation in HIV-infected adults on antiretroviral therapy. Antivir Ther. 2015;20(5):521-7. doi: 10.3851/IMP2940. Epub 2015 Feb 10. PMID 25668820
- [Derived] Funderburg NT, Jiang Y, Debanne SM, Labbato D, Juchnowski S, Ferrari B, Clagett B, Robinson J, Lederman MM, McComsey GA. Rosuvastatin reduces vascular inflammation and T-cell and monocyte activation in HIV-infected subjects on antiretroviral therapy. J Acquir Immune Defic Syndr. 2015 Apr 1;68(4):396-404. doi: 10.1097/QAI.0000000000000478. PMID 25514794
- [Derived] Longenecker CT, Hileman CO, Funderburg NT, McComsey GA. Rosuvastatin preserves renal function and lowers cystatin C in HIV-infected subjects on antiretroviral therapy: the SATURN-HIV trial. Clin Infect Dis. 2014 Oct 15;59(8):1148-56. doi: 10.1093/cid/ciu523. Epub 2014 Jul 11. PMID 25015912
- [Derived] Longenecker CT, Jiang Y, Orringer CE, Gilkeson RC, Debanne S, Funderburg NT, Lederman MM, Storer N, Labbato DE, McComsey GA. Soluble CD14 is independently associated with coronary calcification and extent of subclinical vascular disease in treated HIV infection. AIDS. 2014 Apr 24;28(7):969-77. doi: 10.1097/QAD.0000000000000158. PMID 24691204
- [Derived] Funderburg NT, Jiang Y, Debanne SM, Storer N, Labbato D, Clagett B, Robinson J, Lederman MM, McComsey GA. Rosuvastatin treatment reduces markers of monocyte activation in HIV-infected subjects on antiretroviral therapy. Clin Infect Dis. 2014 Feb;58(4):588-95. doi: 10.1093/cid/cit748. Epub 2013 Nov 18. PMID 24253250
- [Derived] Longenecker CT, Funderburg NT, Jiang Y, Debanne S, Storer N, Labbato DE, Lederman MM, McComsey GA. Markers of inflammation and CD8 T-cell activation, but not monocyte activation, are associated with subclinical carotid artery disease in HIV-infected individuals. HIV Med. 2013 Jul;14(6):385-90. doi: 10.1111/hiv.12013. Epub 2013 Jan 18. PMID 23332012

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rosuvastatin | Sugar Pill Placebo
Started | 72 | 75
Completed | 62 | 57
Not Completed | 10 | 18
Not completed — Lost to Follow-up | 5 | 6
Not completed — Withdrawal by Subject | 3 | 10
Not completed — Adverse Event | 0 | 2
Not completed — Incarcerated | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rosuvastatin | Sugar Pill Placebo | Total
Number analyzed (Participants) | 72 | 75 | 147
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 71 | 75 | 146
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (9) | 45 (10) | 45 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 18 | 32
  Male | 58 | 57 | 115
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 50 | 50 | 100
  White | 20 | 23 | 43
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 72 | 75 | 147
Mean HIV Duration [Mean (Standard Deviation); unit: months] | 140 (79) | 152 (86) | 146 (83)
Mean ARV Duration [Mean (Standard Deviation); unit: months] | 84 (63) | 87 (62) | 86 (62)
Undetectable Viral Load (<48) [Number; unit: participants] | 50 | 56 | 106
Mean Absolute CD4 Count [Mean (Standard Deviation); unit: 10^6 cells/L] | 644 (285) | 636 (312) | 640 (299)

OUTCOME MEASURES:

1. Primary Outcome: Bone Mineral Density (BMD)
Description: Measured by change in bone DEXA from baseline to week 96
Time Frame: 96 weeks
Population: The total number of participants who received this outcome who had valid data is less than the total number of enrolled participants, due to drop outs before week 96 and/or invalid testing data from DEXA results.
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Rosuvastatin | Sugar Pill Placebo
Number analyzed (Participants) | 59 | 55
percentage of change | -0.03 (2.45) | -0.53 (2.70)

2. Primary Outcome: Carotid IMT
Description: changes in carotid IMT is a good measure for cardiovascular disease progression
Time Frame: 96 weeks
Population: The number of participants who received a final CIMT is less than the number of participants enrolled, due in part to study drop outs and/or invalid data measures.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Rosuvastatin | Sugar Pill Placebo
Number analyzed (Participants) | 61 | 55
percentage change | 1.21 (7.97) | 4.04 (9.27)

ADVERSE EVENTS:
Arm/Group | Rosuvastatin | Sugar Pill Placebo
Serious Adverse Events (participants affected / at risk) | 1/72 | 0/75
Other Adverse Events (participants affected / at risk) | 5/72 | 5/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rosuvastatin (N=72) | Sugar Pill Placebo (N=75)
Elevated Creatinine Kinase (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Week 5: Hospitalization secondary to muscle/joint pain; no rhabdomyolysis, no renal compromise. Stopped study drug but remained on study for follow-up.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rosuvastatin (N=72) | Sugar Pill Placebo (N=75)
Elevated Blood Pressure (Cardiac disorders) | 1 (1) | 0 (0)
Muscle, Joint Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) — 2 subjects on placebo reported this AE; no subjects on active drug reported this.
Elevated Glucose (Endocrine disorders) | 0 (0) | 1 (1)
Elevated Creatinine (Renal and urinary disorders) | 1 (1) | 1 (1)
Elevated liver enzymes (Hepatobiliary disorders) | 3 (4) | 2 (2)
Elevated Creatinine Kinase (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No